CLINICAL TRIAL: NCT00806195
Title: A Phase 3b, Open-Label, Randomized, Parallel-Group, Multi-Center Study to Evaluate the Safety of Novartis MenACWY Conjugate Vaccine When Administered With Routine Infant Vaccinations to Healthy Infants
Brief Title: Study to Evaluate the Safety of Novartis MenACWY Conjugate Vaccine When Administered With Routine Infant Vaccinations to Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V59P23
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Results first posted 2013-07-09 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-05

CONDITIONS: Meningitis; Meningococcal Infection
Keywords: vaccine; infants; healthy; meningitis; meningococcal
MeSH Terms: conditions — Meningitis; Meningococcal Infections | interventions — Tetanus Toxoid; Vaccines; Poliovirus Vaccine, Inactivated; Pneumococcal Vaccines; Chickenpox Vaccine; Hepatitis A Vaccines

ARMS (6):
- MenACWY-CRM197 + Routine Vaccines (Non-Detailed) (Experimental): Infants received one vaccination of MenACWY-CRM197 vaccine at 2, 4, 6 and 12 months of age and one vaccination of routine vaccines (according to the local vaccination schedule) - DTaP: 2, 4, 6, 15 months, IPV: 2, 4, 6, months, Hib: 2, 4, 6, 15 months, Pneumococcal conjugate: 2, 4, 6, 12 months, MMR: 12 months.
  Routine vaccines given to subjects in these arms will be consistent with the US ACIP recommended vaccines.
  Non-Detailed - infants who only provided SAEs (Serious Adverse Events) and medically attended AEs (Adverse Events).
  Interventions: Biological: MenACWY-CRM197; Biological: DTaP (Diptheria, Tetanus, Pertussis) Vaccine; Biological: Hib (Haemophilus influenza b) Vaccine; Biological: IPV (Inactivated Polio Vaccine) Vaccine; Biological: Pneumococcal conjugate Vaccine; Biological: MMR (Measles, Mumps, and Rubella) Vaccine
- Routine Vaccines (Non-Detailed) (Active Comparator): Infants received one vaccination of routine vaccines (according to the local vaccination schedule) - DTaP: 2, 4, 6, 15 months, IPV: 2, 4, 6 months, Hib: 2, 4, 6, 15 months, Pneumococcal conjugate: 2, 4, 6, 12 months, MMR: 12 months.
  Routine vaccines given to subjects in these arms will be consistent with the US ACIP recommended vaccines.
  Non-Detailed - subjects who only provided SAEs and medically attended AEs.
  Interventions: Biological: DTaP (Diptheria, Tetanus, Pertussis) Vaccine; Biological: Hib (Haemophilus influenza b) Vaccine; Biological: IPV (Inactivated Polio Vaccine) Vaccine; Biological: Pneumococcal conjugate Vaccine; Biological: MMR (Measles, Mumps, and Rubella) Vaccine
- MenACWY-CRM197 + Routine Vaccines (Detailed) (Experimental): Infants received one vaccination of MenACWY-CRM197 vaccine at 2, 4, 6 and 12 months of age and one vaccination of routine vaccines (according to the local vaccination schedule) - DTaP: 2, 4, 6, 15 months, IPV: 2, 4, 6, months, Hib: 2, 4, 6, 15 months, Pneumococcal conjugate: 2, 4, 6, 12 months, MMR, Varicella, Hepatitis A: 12 months. HBV and rotavirus vaccines should be administered according to ACIP guidelines during the first year of life.
  Routine vaccines given to subjects in these arms will be consistent with the US ACIP recommended vaccines.
  Detailed - subjects who provided Reactogenicity and all AEs for 7 days, SAEs and medically attended AEs.
  Interventions: Biological: MenACWY-CRM197; Biological: DTaP (Diptheria, Tetanus, Pertussis) Vaccine; Biological: Hib (Haemophilus influenza b) Vaccine; Biological: IPV (Inactivated Polio Vaccine) Vaccine; Biological: Pneumococcal conjugate Vaccine; Biological: MMR (Measles, Mumps, and Rubella) Vaccine; Biological: Varicella Vaccine; Biological: Hepatitis A Virus
- Routine Vaccines (Detailed) (Active Comparator): Infants received one vaccination of routine vaccines (according to the local vaccination schedule) - DTaP: 2, 4, 6, 15 months, IPV: 2, 4, 6 months, Hib: 2, 4, 6, 15 months, Pneumococcal conjugate: 2, 4, 6, 12 months, MMR, Varicella, and Hepatitis A: 12 months. HBV and rotavirus vaccines should be administered according to ACIP guidelines during the first year of life.
  Routine vaccines given to subjects in these arms will be consistent with the US ACIP recommended vaccines.
  Detailed - subjects who provided Reactogenicity and all AEs for 7 days, SAEs and medically attended AEs.
  Interventions: Biological: DTaP (Diptheria, Tetanus, Pertussis) Vaccine; Biological: Hib (Haemophilus influenza b) Vaccine; Biological: IPV (Inactivated Polio Vaccine) Vaccine; Biological: Pneumococcal conjugate Vaccine; Biological: MMR (Measles, Mumps, and Rubella) Vaccine; Biological: Varicella Vaccine; Biological: Hepatitis A Virus
- MenACWY-CRM197 + Routine Vaccines (All) (Experimental): Infants received one vaccination of MenACWY-CRM197 vaccine at 2, 4, 6 and 12 months of age and one vaccination of routine vaccines (according to the local vaccination schedule) - DTaP: 2, 4, 6, 15 months, IPV: 2, 4, 6, months, Hib: 2, 4, 6, 15 months, Pneumococcal conjugate: 2, 4, 6, 12 months, MMR, Varicella, Hepatitis A: 12 months. HBV and rotavirus vaccines should be administered according to ACIP guidelines during the first year of life.
  Routine vaccines given to subjects in these arms will be consistent with the US ACIP recommended vaccines.
  All (Detailed and Non-Detailed subjects): Detailed - subjects who provided Reactogenicity and all AEs for 7 days, SAEs and medically attended AEs; Non-Detailed - subjects who only provided SAEs and medically attended AEs.
  Interventions: Biological: MenACWY-CRM197; Biological: DTaP (Diptheria, Tetanus, Pertussis) Vaccine; Biological: Hib (Haemophilus influenza b) Vaccine; Biological: IPV (Inactivated Polio Vaccine) Vaccine; Biological: Pneumococcal conjugate Vaccine; Biological: MMR (Measles, Mumps, and Rubella) Vaccine; Biological: Varicella Vaccine; Biological: Hepatitis A Virus
- Routine Vaccines (All) (Active Comparator): Infants received one vaccination of routine vaccines (according to the local vaccination schedule) - DTaP: 2, 4, 6, 15 months, IPV: 2, 4, 6, months, Hib: 2, 4, 6, 15 months, Pneumococcal conjugate: 2, 4, 6, 12 months, MMR, Varicella, and Hepatitis A: 12 months. HBV and rotavirus vaccines should be administered according to ACIP guidelines during the first year of life.
  Routine vaccines given to subjects in these arms will be consistent with the US ACIP recommended vaccines.
  All (Detailed and Non-Detailed subjects): Detailed - subjects who provided Reactogenicity and all AEs for 7 days, SAEs and medically attended AEs; Non-Detailed - subjects who only provided SAEs and medically attended AEs.
  Interventions: Biological: DTaP (Diptheria, Tetanus, Pertussis) Vaccine; Biological: Hib (Haemophilus influenza b) Vaccine; Biological: IPV (Inactivated Polio Vaccine) Vaccine; Biological: Pneumococcal conjugate Vaccine; Biological: MMR (Measles, Mumps, and Rubella) Vaccine; Biological: Varicella Vaccine; Biological: Hepatitis A Virus

INTERVENTIONS:
Biological: MenACWY-CRM197 — Four 0.5mL vaccinations of MenACWY-CRM197 conjugate vaccine was administered by intramuscular injection at 2, 4, 6 and 12 months of age.
  Arms: MenACWY-CRM197 + Routine Vaccines (All); MenACWY-CRM197 + Routine Vaccines (Detailed); MenACWY-CRM197 + Routine Vaccines (Non-Detailed)
Biological: DTaP (Diptheria, Tetanus, Pertussis) Vaccine — Four vaccinations of DTaP (Diptheria, Tetanus, Pertussis) was administered at 2, 4, 6, and 15 months of age.
Biological: Hib (Haemophilus influenza b) Vaccine — Four vaccinations of Hib (Haemophilus influenza b) vaccine was administered at 2, 4, 6 and 15 months of age.
Biological: IPV (Inactivated Polio Vaccine) Vaccine — Three vaccinations of IPV (Inactivated Polio Vaccine) was administered at 2, 4, and 6 months of age.
Biological: Pneumococcal conjugate Vaccine — Four vaccinations of Pneumococcal conjugate vaccine was administered at 2, 4, 6 and 12 months of age.
Biological: MMR (Measles, Mumps, and Rubella) Vaccine — One vaccination of MMR (Measles, Mumps, and Rubella) was administered at 12 months of age.
Biological: Varicella Vaccine — One vaccination of Varicella vaccine was administered at 12 months of age.
  Arms: MenACWY-CRM197 + Routine Vaccines (All); MenACWY-CRM197 + Routine Vaccines (Detailed); Routine Vaccines (All); Routine Vaccines (Detailed)
Biological: Hepatitis A Virus — One vaccination of Hepatitis A Virus vaccine was administered at 12 months of age.
  Arms: MenACWY-CRM197 + Routine Vaccines (All); MenACWY-CRM197 + Routine Vaccines (Detailed); Routine Vaccines (All); Routine Vaccines (Detailed)

SUMMARY:
The primary objective of this phase 3b study is to evaluate the safety and tolerability of Novartis MenACWY conjugate vaccine when administered with routine infant vaccinations to healthy infants

ELIGIBILITY:
Inclusion Criteria:

* healthy 2-month-old infants (aged 55 - 89 days); babies must have been born after a full-term pregnancy with an estimated gestation age ≥37 weeks and a birth weight ≥2.5 kg
* for whom a parent/legal representative has given written informed consent after the nature of the study has been explained;
* who are available for all visits scheduled in the study;
* who are in good health as determined by medical history and physical assessment.

Exclusion Criteria:

* who previously received any meningococcal vaccine or D, T, P, IPV or OPV, H influenzae type b (Hib) or Pneumococcus; prior doses of BCG (one) and/or HBV (two) are permitted
* who have a previous confirmed or suspected disease caused by N meningitidis, C diphtheriae, C tetani, Poliovirus, Hepatitis B, Hib, Pneumococcus or B pertussis (history of laboratory confirmed, or clinical condition of paroxysmal cough for a period of longer than or equal to 2 weeks associated with apnea or whooping);
* who have had household contact with and/or intimate exposure to an individual with laboratory confirmed N meningitidis (serogroups A, C, W135, or Y), B pertussis, Hib, C diphtheriae, Polio, or pneumococcal infection at any time since birth;
* who have a history of anaphylactic shock, asthma, urticaria or other allergic reaction after previous vaccinations or known hypersensitivity to any vaccine component;
* who have experienced significant acute or chronic infection within the previous 7 days or have experienced fever (axillary temperature ≥ 38.0°C [100.4°F]) within the previous 3 days;
* who have any present or suspected serious acute (e.g. leukemia, lymphomas), or chronic disease (e.g., with signs of cardiac disease, renal failure, severe malnutrition, or insulin dependent diabetes), or progressive neurological disease, or a genetic anomaly/known cytogenic disorders (e.g., Down's syndrome);
* who have a known or suspected autoimmune disease or persistent impairment/alteration of immune function resulting from (for example):

  1. receipt of any immunosuppressive therapy at any time since birth
  2. receipt of immunostimulants at any time since birth
  3. receipt of any systemic corticosteroid since birth;
* who have a suspected or known HIV infection or HIV related disease;
* who have ever received blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation;
* who have a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time;
* who have any history of seizure;
* who with their parents/legal representatives are planning to leave the area of the study site before the end of the study period;
* who have any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives;
* who have received any investigational agents or vaccines since birth or who expect to receive an investigational agent or vaccine prior to the completion of the study.
* who are relatives of site research staff working on this study.

Ages: 55 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7744 (Actual)
Dates: Start 2008-12; Primary Completion 2011-03 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (153):
- United States (130):
  - 6 Alabama Clinical Therapeutics 806 St. Vincent's Drive, Ste 615, Birmingham, Alabama
  - 43 Alabama Clinical Therapeutics, LLC 364 Honeysuckle Rd, Dothan, Alabama
  - 81 Cholla Pediatrics 2167 West Orange Grove Road, Tuscon, Arizona
  - 55 Central Arkansas Pediatric Clinic Pediatric 2301 Springhill Road Suite 200, Benton, Arkansas
  - 21 Northwest Arkansas Pediatric Clinic 3383 N. MANA Court Suite 101, Fayetteville, Arkansas
  - 30 Sparks Pediatric Clinic 1501 S. Waldron Road Suite 100, Fort Smith, Arkansas
  - 14 The Children's Clinic of Jonesboro 800 S. Church Suite 400, Jonesboro, Arkansas
  - 170 Little Rock Children's Clinic P.A. 9600 Lile Dr., Ste 360, Little Rock, Arkansas
  - 3 Arkansas Pediatric Clinic 500 S. University Suite 200, Little Rock, Arkansas
  - 179 Associated Pharmaceutical Research Center, Inc 8615 Knott Avenue Suite 5, Buena Park, California
  - 160 San Fernando Valley Research Associates, Inc. 7111 Winnetka Ave. #14, Canoga Park, California
  - 157 Universal Biopharma Research Institute Inc./Alta Family Health Clinic 888 N. Alta Ave., Dinuba, California
  - 1 Premier Health Research Center, LLC 11525 Brookshire Ave Suite 400, Downey, California
  - 68 Sierra Medical Research 5150 N. Sixth, Suite 156, Fresno, California
  - 129 Citrus Vally Family Practice 1400 Hacienda Blvd, La Puente, California
  - 114 Loma Linda University Health 11175 Campus Street Coleman Pavillion A-1120, Loma Linda, California
  - 59 Loma Linda University Health 11175 Campus Street Coleman Pavillion A-1120, Loma Linda, California
  - 153 Health Care Partners Medical Group Health Care Partners Medical Group 4401 Atlantic Ave., Long Beach, California
  - 94 Health Care Partners Medical Group 1025 W. Olympic Blvd., Los Angeles, California
  - 67 Madera Family Medical Group 1111 West 4th Street, Madera, California
  - 121 Kaiser Permanente (Oakland) 3505 Broadway 6th floor, Oakland, California
  - 63 Kaiser Permanente Vaccine Study Center One Kaiser Plaza 16th Floor, Oakland, California
  - 42 Children's Hospital of Orange County 455 S. Main Street, Orange, California
  - 12 Center For Clinical Trials, LLC. 16660 Paramount Blvd Suite 301, Paramount, California
  - 122 Kaiser Permanente (Pleasanton) 7601 Stoneridge Drive, MOB North 2nd Floor, Pleasanton, California
  - 57 UC Davis Medical Center 2516 Stockton Blvd Ticon II, Sacramento, California
  - 123 Kaiser Permanente (San Francisco) 2200 O'Farrell Street 6th floor room 636, San Francisco, California
  - 166 Buena Salud Pediatrics 2880 Story Road, San Jose, California
  - 20 White Memorial Pediatric Medical Group UCLA Center for Vaccine Research 1124 West Carson Street Liu Research Building (Room 132), Torrance, California
  - 152 Health Care Partners Medical Group 3565 Del Amo Blvd Research Dept., Torrance, California
  - 40 Center for Clinical Trials of San Gabriel 1300 S Sunset Avenue Suite 101, West Covina, California
  - 54 1st International Research Centers 10370 Steeke Street, Thornton, Colorado
  - 29 Norwich Pediatric Group 92 New London Turnpike, Norwich, Connecticut
  - 99 Altamonte Pediatric Associates 101 N Country Club Rd., Lake Mary, Florida
  - 60 Orlando Health Pediatric Faculty Practice 32 West Sturtevant St, MP-141, Orlando, Florida
  - 34 Pediatric Partners Pediatrics 3401 PGA Blvd Ste 300, Palm Beach Gardens, Florida
  - 88 Physician Care Clinical Research 1918 Robinhood Street, Sarasota, Florida
  - 162 North Georgia Clinical Research Center 1575 Chattanooga Avenue Suite 1, Dalton, Georgia
  - 11 Pediatrics and Adolescent Medicine, PA 2155 Post Oak Tritt Road Suite 100, Marietta, Georgia
  - 101 Pediatrics and Adolescent Medicine, PA 120 Stonebridge Parkway, Suite 410, Woodstock, Georgia
  - 132 Kaiser Permanente Pediatric - Mapunapuna 2828 Paa Street, 2nd Floor, Honolulu, Hawaii
  - 131 Kaiser Permanente Waipio 1st Floor 94-1480 Moaniani Street, Waipahu, Hawaii
  - Northern Illinois Research Associates 625 E. Bethany Ste. 3, DeKalb, Illinois
  - 95 Heartland Research Associates 510 West Radio Lane, Arkansas City, Kansas
  - 92 Heartland Research Associates LLC 700 Medical Center Dr. Suite 210, Newton, Kansas
  - 178 Pediatric Care 6725 Southwest Twenty-Ninth Street, Topeka, Kansas
  - 51 Kentucky Pediatric/Adult Research 201 S. 5th Street, Bardstown, Kentucky
  - 84 Michael W. Simon M.D. 185 Pasadena Drive Suite 220, Lexington, Kentucky
  - 106 University Child Health Specialists 230 East Broadway, Louisville, Kentucky
  - 24 Bluegrass Clinical Research, Inc 5512 Bardstown Road Suite 2, Louisville, Kentucky
  - 76 Bluegrass Clinical Research, Inc 5512 Bardstown Road Suite2, Louisville, Kentucky
  - 15 University of Louisville 571 South Floyd Suite 321 L, Ouisville, Kentucky
  - 108 Physicians to Children and Adolescents 102 West Depot Street, Springfield, Kentucky
  - 86 Willis-Knighton Physician Network 7847 Youree Drive, Shreveport, Louisiana
  - 22 Roslindale Pediatric Assoc, P.C 1153 Centre St Suite 31, Boston, Massachusetts
  - 23 Pediatric Associates of Fall River 829 South Main Street, Fall River, Massachusetts
  - 126 North Andover Pediatrics Associates 800 Turnpike Street, North Andover, Massachusetts
  - 9 Woburn Pediatric Associates 7 Alfred Street Baldwin Park II, Woburn, Massachusetts
  - 168 Southwestern Medical Clinic 2002 South 11th Street, Niles, Michigan
  - 26 Southwestern Medical Clinic 5515 Cleveland Avenue Suite 1, Stevensville, Michigan
  - 89 Aspen Medical Group 1020 Bandana Blvd West Ste 214, Saint Paul, Minnesota
  - 80 Craig A. Spiegel, M.D 12255 DePaul Drive Sutie 380, Bridgeton, Missouri
  - 69 Clinical Research Center of Nevada 1012 East Sahara Avenue, Las Vegas, Nevada
  - 173 Maimonides Medical Center 948 48th Street 1st Floor, Brooklyn, New York
  - 70 Summer Pediatrics 4811 Buckley Road, Liverpool, New York
  - 16 Winthrop University Hospital Department of Pediatrics 120 Mineola Blvd Suite 210, Mineola, New York
  - 77 SUNY Upstate Medical University 750 East Adams Street Suite 5400, Syracuse, New York
  - 56 Cary Pediatrics 1001 Crescent Green Dr., Cary, North Carolina
  - 103 Durham Pediatrics 2609 North Duke Street, Suite 1000, Durham, North Carolina
  - 104 Regional Pediatrics 4022 Freedom Lake Drive, Durham, North Carolina
  - 13 Duke Health Center 4020 N. Roxboro Road, Durham, North Carolina
  - 48 Capitol Pediatrics and Adolescent Center 3801 Computer Drive Suite 200, Raleigh, North Carolina
  - 91 Triangle Medical Research 5816 Creedmoor Rd. Suite 104, Raleigh, North Carolina
  - 73 Piedmont Medical Research Assoc 1901 S Hawthorne Rd Ste 306, Winston-Salem, North Carolina
  - 87 Innovis Health 1702 South University Drive Suite 1, Fargo, North Dakota
  - 97 Children's Hospital Medical Center of Akron One Perkins Square, Akron, Ohio
  - 120 Akron Children's Hospital Pediatrics 62 Conservatory Drive, #A, Barberton, Ohio
  - 36 Dr. Senders and Associates, Pediatrics 2054 South Green Road, Cleveland, Ohio
  - 79 Dayton Clinical Research 1100 Salem Ave, Dayton, Ohio
  - 37 Pediatric Associates of Fairfield, Inc. 5900 Boymel Drive, Fairfield, Ohio
  - 4 Ohio Pediatrics, INC 7371 Brandt Pike Suite C, Huber Heights, Ohio
  - 102 Ohio Pediatrics, INC 1775 Delco Park Drive, Kettering, Ohio
  - 28 Pediatric Associates of Youngstown 4308 Belmont Avenue, Youngstown, Ohio
  - 100 Pediatric Associates of Youngstown 727 East Western Reserve Road, Youngstown, Ohio
  - 25 Oklahoma State University-CHS C/O Pediatrics 635 West 11th Street, Tulsa, Oklahoma
  - 83 The Portland Clinic LLP 15950 SW Millikan Lane Research Dept., Beaverton, Oregon
  - 7 Cyn3rgy Research 24850 SE Stark Street Suite 180, Gresham, Oregon
  - 113 Children's Health Care-West 4671 West Lake Road, Erie, Pennsylvania
  - 109 UPMC/Community Medicine Inc. 90 Shenango Street, Greenville, Pennsylvania
  - 107 Pennridge Pediatric Associates 270 Main Street, Harleysville, Pennsylvania
  - 110 Pediatric Alliance Southwestern - Squirrel Hill 4070 Beechwood Blvd, Pittsburgh, Pennsylvania
  - 112 Pediatric Alliance, Southwestern 850 Clairton Blvd, Pittsburgh, Pennsylvania
  - 118 Pediatric Alliance, PC Arcadia Division 9000 Perry Highway Suite 120, Pittsburgh, Pennsylvania
  - 5 Primary Physicians Research, Inc 1580 McLaughlin Run Road, Pittsburgh, Pennsylvania
  - 49 Pennridge Pediatric Associates 711 Lawn Avenue, Sellersville, Pennsylvania
  - 41 Palmetto Pediatrics, PA Pediatrics 2781 Tricom Street, Charleston, South Carolina
  - 71 Holston Medical Group 105 W. Stone Dr. Suite 2A, Kingsport, Tennessee
  - 72 Holston Medical Group 2033 Meadowview Lane, Kingsport, Tennessee
  - 165 Focus Research Group 201 Signature Place Suite C, Lebanon, Tennessee
  - 52 Heritage Medical Associates 2325 Crestmoor Road, Nashville, Tennessee
  - 90 Premier Medical Group Alpha Clinical Research 279 Clear Sky Court, Ste C Clarksville, Tennessee
  - 64 Amarillo Childrens Clinical Research #17 Care Circle, Amarillo, Texas
  - 19 University of North Texas Health Science Center 3500 Camp Bowie Blvd, Fort Worth, Texas
  - 175 Sealy Center for Vaccine Development, Clinical Trials 301 University Blvd. Children's Hospital Room 3.270F L#20412, Galveston, Texas
  - 96 West Houston Clinical Research Service 2026 Wirt Road, Houston, Texas
  - 50 San Antonio Metropolitan Health District 332 West Commerce Room 307, San Antonio, Texas
  - 31 Southwest Children's Research Associates, P. A. 5282 Medical Drive Suite 311, San Antonio, Texas
  - 47 Dynamed Clinical Research 13406 Medical Complex Dr Suite 200, Tomball, Texas
  - 75 Pediatric Care 1596 S. 500 W., 1st Floor, Bountiful, Utah
  - 82 Dixie Pediatrics 1240 E 100 S STE 14 St., George, Utah
  - 115 Wee Care(Layton) 1580 West Antelope Drive, Layton, Utah
  - 116 Wee Care(Kaysville) 934 South Main Street, Suite 8, Layton, Utah
  - 181 Jean Brown Research 164 East 5900 South Suite A-112, Murray, Utah
  - 74 Utah Valley Pediatrics North University 7407 North Cedar St., Provo, Utah
  - 117 Wee Care(Roy) 5991 South 3500 West, Suite 100, Roy, Utah
  - 66 J. Lewis Research Inc. 2295 Foothill Drive, Salt Lake City, Utah
  - 61 Foothill Family Clinic South 6360 South 300 East Suite 100, Salt Lake City, Utah
  - 151 Family First Pediatrics c/o Pharmaceutical Research Organization 1268 W. South Jordan Parkway Suite 201, South Jordan, Utah
  - 44 Wee Care Pediatrics (Syracuse) 1792 West 1700 South Suite 102, Syracuse, Utah
  - Jordan Ridge Kids & Teens 8822 S. Redwood Road Suite S103, West Jordan, Utah
  - 85 Pediatric Research of Charlottesville, LLC 1011 East Jefferson St. Suite 3, Charlottesville, Virginia
  - 158 Huguenot Pediatrics, PC 1407 Huguenot Rd., Midlothian, Virginia
  - 46 Virginia Commonwealth University 1001 East Marshall Street P008, Richmond, Virginia
  - 93 Advanced Pediatrics 100 East Street SE Suite 301, Vienna, Virginia
  - 2 Rockwood Clinical Research Center 400 East Fifth Avenue, Spokane, Washington
  - 38 Rockwood Clinic, P.S. 9001 N. Country Homes Blvd., Spokane, Washington
  - 124 The Vancouver Clinic/NE 87th Avenue 700 NE 87th Avenue, Vancouver, Washington
  - 125 The Vancouver Clinic/Columbia Tech Center 501 SE 172th Avenue, Vancouver, Washington
  - 167 The Vancouver Clinic/Salmon Creek 2525 NE 139th Street, Vancouver, Washington
  - 163 Wenatchee Valley Medical Center Clinical Research Department 820 North Chelan Avenue, Wenatchee, Washington
- China (4):
  - 304 Department of Pediatrics, Chang Gung Children's Hospital 12F, L Building, #5, Fu-Shin St., Kweishan, Taoyuan 333, Taiwan
  - 301 Department of Pediatrics, National Taiwan University Hospital, 15F,Children's Hospital, No. 8 Chung Shan S. Rd,, Taipei, Taiwan
  - 302 Department of Pediatrics, Mackay Memorial Hospital No. 92, Sec. 2, ChangShan Road,, Taipei, Taiwan
  - 303 Department of Pediatrics, Taiwan Adventist Hospital 424, Sec 2, Pa-Te Road,, Taipei, Taiwan
- Costa Rica (4):
  - 401 Clínica Pediátrica Calle 20 Ave 0 y 2 Costado Oeste del Hospital Nacional de Niños - segundo piso,, San José, Costa Rica
  - 402 Centro Integral Medico 25 m Oeste e la Junta de Protección Social,, San José, Costa Rica
  - 404 Instituto de Atención Pediátrica (IAP) Del Restaurante La Bastilla, 50m Sur, Paseo Colón, San José, Costa Rica
  - 403 Centro Médico San Vicente 125m Este de la entrada Principal de Emergencia del Hospital, San Vicente de Paul, Heredia, Costa Rica
- Guatemala (7):
  - 501 Hospital Infantil de Infectología y Rehabilitación 9ª. Avenida 7-01 Zona 11 Colonia Roosevelt,, Guatemala City, Departamento de Guatemala
  - 507 Clínica Médica Privada Edificio Multimédica, 2 calle 25-19 Zona 15, Vista Hermosa I, Guatemala CP 01015
  - 508 Unidad de Crecimiento y Desarrollo, Clínica del Niño Sano, Hospital Roosevelt 6ª Avenida 3-10 Zona 11, Ingreso Principal Hospital Roosevelt, Guatemala City, Guatemala CP. 01011
  - 502 Clínica Privada 6a Avenida 3-22 Zona 10, Centro Médico II, Ofic. 601, Guatemala City, Guatemala Cp01010
  - 503 Clínica para Niños 6a Avenida 6-63 Zona 10, Edificio Sixtino, Oficina 305, Tercer Nivel,, Guatemala City, Guatemala Cp01010
  - 506 Health Center 4ª Avenida 16-72 Zona 10,, Guatemala City, Guatemala Cp01010
  - 504 Clínica Periférica El Amparo II, 38 Calle 31-89, Zona 7 Colonia El Amparo II,, Guatemala City, Guatemala. CP 01007
- Panama (3):
  - 601 Hospital Materno Infantil José Domingo De Obaldía, Centro para la Investigación y Desarrollo de Estudios Clínicos Vía Panamericana, San Pablo viejo, David,, Chiriquí
  - 602 Centro Pediátrico América, Consultorio América Segundo Piso Consultorio No. 223, Vía España, Carrasquilla, Frente al Hospital de Especialidades Pediátricas, Panama City
  - 603 Policentro Luis H. Moreno, Parque Lefevre, Via Cincuentenario
- Peru (5):
  - 704 Hospital Nacional Docente Madre Niño San Bartolomé Av. Alfonso Ugarte 825,, Lima Cercado, Lima 01
  - 701 Instituto de Investigación Nutricional - Anexo Huáscar, SJL Manzana 122, Lote 21, Grupo 15, Huascar, San Juan de Lurigancho, Lima 36
  - 703 Hospital María Auxiliadora Av. Miguel Iglesias 968, San Juan de Miraflores,, Lima
  - 705 Hospital Nacional Cayetano Heredia Av. Honorio Delgado No. 262, Urbanización Ingeniería, San Martín de Porres, Lima
  - 708 Hospital Nacional Guillermo Almenara Irigoyen Av. Grau No. 800, La Victoria, Lima 13, Lima

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects enrolled were included in the trial.
Groups:
- MenACWY-CRM197 + Routine Vaccines (Non-detailed): Infants received one vaccination of MenACWY-CRM197 vaccine at 2, 4, 6 and 12 months of age and one vaccination of routine vaccines (according to the local vaccination schedule) - DTaP: 2, 4, 6, 15 months, IPV: 2, 4, 6, months, Hib: 2, 4, 6, 15 months, Pneumococcal conjugate: 2, 4, 6, 12 months, MMR: 12 months.
  Routine vaccines given to subjects in these arms will be consistent with the US ACIP recommended vaccines.
  Non-Detailed - subjects who only provided Serious Adverse Events (SAEs) and medically attended Adverse (AE).
- Routine Vaccines (Detailed): Infants received one vaccination of routine vaccines (according to the local vaccination schedule) - DTaP: 2, 4, 6, 15 months, IPV: 2, 4, 6 months, Hib: 2, 4, 6, 15 months, Pneumococcal conjugate: 2, 4, 6, 12 months, MMR, Varicella, and Hepatitis A: 12 months. HBV and rotavirus vaccines should be administered according to ACIP guidelines during the first year of life.
  Routine vaccines given to subjects in these arms will be consistent with the US ACIP recommended vaccines.
  Detailed - subjects who provided Reactogenicity, all AEs for 7 days, SAEs and medically attended AEs.
Period: Overall Study
Arm/Group | MenACWY-CRM197 + Routine Vaccines (Non-detailed) | Routine Vaccines (Non-detailed) | MenACWY-CRM197 + Routine Vaccines (Detailed) | Routine Vaccines (Detailed)
Started | 4363 | 1483 | 1409 | 489
Completed | 3849 | 1321 | 1139 | 383
Not Completed | 514 | 162 | 270 | 106
Not completed — Death | 6 | 0 | 1 | 0
Not completed — Adverse Event | 25 | 5 | 11 | 2
Not completed — Withdrawal by Subject | 119 | 31 | 76 | 35
Not completed — Lost to Follow-up | 217 | 66 | 90 | 34
Not completed — Inappropriate Enrollment | 0 | 1 | 0 | 0
Not completed — Administrative Reason | 113 | 35 | 66 | 26
Not completed — Protocol Violation | 34 | 24 | 26 | 9

BASELINE CHARACTERISTICS:
Groups:
- MenACWY-CRM197 + Routine Vaccines (Non-Detailed): Infants received one vaccination of MenACWY-CRM197 vaccine at 2, 4, 6 and 12 months of age and one vaccination of routine vaccines (according to the local vaccination schedule) - DTaP: 2, 4, 6, 15 months, IPV: 2, 4, 6, months, Hib: 2, 4, 6, 15 months, Pneumococcal conjugate: 2, 4, 6, 12 months, MMR: 12 months.
  Routine vaccines given to subjects in these arms will be consistent with the US ACIP recommended vaccines.
  Non-Detailed - subjects who only provided SAEs and medically attended AEs.
- Total: Total of all reporting groups
Arm/Group | MenACWY-CRM197 + Routine Vaccines (Non-Detailed) | Routine Vaccines (Non-Detailed) | MenACWY-CRM197 + Routine Vaccines (Detailed) | Routine Vaccines (Detailed) | Total
Number analyzed (Participants) | 4363 | 1483 | 1409 | 489 | 7744
Age Continuous [Mean (Standard Deviation); unit: Days] | 64.9 (7.4) | 64.7 (7.1) | 65.5 (6.5) | 65.2 (6.3) | 65.0 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2135 | 703 | 716 | 232 | 3786
  Male | 2228 | 780 | 693 | 257 | 3958

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With At Least One Severe Systemic Reaction After Any Vaccination
Description: To compare the percentages of subjects who reported at least one severe systemic reaction after any vaccination of MenACWY-CRM197 (detailed) plus routine vaccines (detailed) group to that observed in the routine vaccines alone (detailed) group administered at 2, 4, 6, and 12 months of age.
  Detailed - infants who provided reactogenicity and all Adverse Events (AEs) for 7 days, Serious Adverse Events (SAEs) and medically attended AEs.
Time Frame: 15 minutes to Day 7 after any vaccination administered at 2, 4, 6 and 12 months of age
Population: Analysis was done on As Treated Safety Population - Subjects who received at least one study dose and provided postbaseline safety data, and that subjects would be included in the group for the vaccination actually received (i.e., analyzed as treated).
Measure: Number; unit: Percentages of subjects
Groups:
- MenACWY-CRM197 + Routine Vaccines (Detailed): Infants received one vaccination of MenACWY-CRM197 vaccine at 2, 4, 6 and 12 months of age and one vaccination of routine vaccines (according to the local vaccination schedule) - DTaP: 2, 4, 6, 15 months, IPV: 2, 4, 6, months, Hib: 2, 4, 6, 15 months, Pneumococcal conjugate: 2, 4, 6, 12 months, MMR, Varicella, Hepatitis A: 12 months. HBV and rotavirus vaccines should be administered according to ACIP guidelines during the first year of life.
  Routine vaccines given to subjects in these arms will be consistent with the US ACIP recommended vaccines.
  Detailed - infants who provided reactogenicity and all Adverse Events (AEs) for 7 days, Serious Adverse Events (SAEs) and medically attended AEs.
- Routine Vaccines (Detailed): Infants received one vaccination of routine vaccines (according to the local vaccination schedule) - DTaP: 2, 4, 6, 15 months, IPV: 2, 4, 6 months, Hib: 2, 4, 6, 15 months, Pneumococcal conjugate: 2, 4, 6, 12 months, MMR, Varicella, and Hepatitis A: 12 months. HBV and rotavirus vaccines should be administered according to ACIP guidelines during the first year of life.
  Routine vaccines given to subjects in these arms will be consistent with the US ACIP recommended vaccines.
  Detailed - infants who provided reactogenicity and all Adverse Events (AEs) for 7 days, Serious Adverse Events (SAEs) and medically attended AEs.
Arm/Group | MenACWY-CRM197 + Routine Vaccines (Detailed) | Routine Vaccines (Detailed)
Number analyzed (Participants) | 1349 | 461
Percentages of subjects | 16 | 13
Statistical Analysis 1: Comparison: MenACWY-CRM197 + Routine Vaccines (Detailed) vs Routine Vaccines (Detailed); MenACWY-CRM 197 administered concomitantly with routine vaccines was considered noninferior to routine vaccines alone with respect to severe systemic reactions if the upper limit of the 2-sided 95% CI of the difference (MenACWY-CRM197 vaccine plus routine vaccines group minus routine vaccines only group) in the proportion of subjects experiencing at least one severe systemic reaction during the first 7 days (days 1-7) after any vaccination was <6%; Test type: Non-Inferiority or Equivalence — The null hypothesis associated with the safety objective was that the upper limit of the two-sided 95% CI for this difference in the proportion of subjects experiencing at least one severe systemic reaction during the first 7 days after any vaccination (PMenACWY+Routine Vaccines-PRoutine Vaccines) was ≥ 6%; Miettinen and Nurminen; Mean Difference (Final Values) = 3.0, 95% CI 2-sided [-0.8 to 6.4]

2. Secondary Outcome: Percentages of Subjects With At Least One Serious Adverse Event During the Entire Study Period
Description: To compare the percentages of subjects presenting at least one serious adverse event (SAE) through 6 months post-final dose in subjects who received MenACWY-CRM197 vaccine concomitantly with routine vaccinations to the percentages of subjects who received routine vaccinations alone.
Time Frame: Day 1 (2 months of age) to 18 months of age
Population: Analysis was done on as treated safety population.
Measure: Number; unit: Percentages of subjects
Arm/Group | MenACWY-CRM197 + Routine Vaccines (All) | Routine Vaccines (All)
Number analyzed (Participants) | 5760 | 1968
Percentages of subjects | 6 | 6
Statistical Analysis 1: Comparison: MenACWY-CRM197 + Routine Vaccines (All) vs Routine Vaccines (All); MenACWY-CRM 197 administered concomitantly with routine vaccines was considered non inferior to routine vaccines alone with respect to serious adverse events if the upper limit of the 2-sided 95% CI of the difference (MenACWY vaccine plus routine vaccines group minus routine vaccines only group) of the proportion of subjects experiencing at least one serious adverse event was <5%; Test type: Non-Inferiority or Equivalence — The null hypothesis associated with the SAE safety objective was that the upper limit of the two-sided 95% confidence interval for the difference between the MenACWY and routine vaccine groups in the proportion of subjects experiencing at least one SAE (PMenACWY + Routine Vaccines - PRoutine Vaccines) was ≥5%; Miettinen and Nurminen; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.9 to 1.5]
Statistical Analysis 2: Comparison: MenACWY-CRM197 + Routine Vaccines (All) vs Routine Vaccines (All); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — The null hypothesis associated with the SAE safety objective was that the upper limit of the two-sided 95% confidence interval for the difference between the MenACWY and routine vaccine groups in the proportion of subjects experiencing at least one SAE (PMenACWY + Routine Vaccines - PRoutine Vaccines) was <5%; Miettinen and Nurminen; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.8 to 1.3]

3. Secondary Outcome: Percentages of Subjects Reporting Solicited Adverse Events, After Each Vaccination
Description: To compare the percentage of subjects who reported local and systemic solicited adverse events from day 1 to day 7 after each vaccination with MenACWY-CRM197 given concomitantly with routine vaccinations to the routine vaccinations alone group.
Time Frame: 15 minutes to Day 7
Population: Analysis was done on as treated safety population.
Measure: Number; unit: percentages of subjects
Groups:
- MenACWY-CRM 197 + Routine Vaccines (Detailed): Infants received one vaccination of MenACWY-CRM197 vaccine at 2, 4, 6 and 12 months of age and one vaccination of routine vaccines (according to the local vaccination schedule) - DTaP: 2, 4, 6, 15 months, IPV: 2, 4, 6, months, Hib: 2, 4, 6, 15 months, Pneumococcal conjugate: 2, 4, 6, 12 months, MMR, Varicella, Hepatitis A: 12 months. HBV and rotavirus vaccines should be administered according to ACIP guidelines during the first year of life.
  Routine vaccines given to subjects in these arms will be consistent with the US ACIP recommended vaccines.
  Detailed - subjects who provided reactogenicity and all AEs for 7 days, SAEs and medically attended AEs.
Arm/Group | MenACWY-CRM 197 + Routine Vaccines (Detailed) | Routine Vaccines (Detailed)
Number analyzed (Participants) | 1313 | 451
percentages of subjects
  Any Local (2 month vaccination) (N=1313, 451) | 53 | 56
  Injection Site Tenderness (N=1301, 446) | 46 | 49
  Injection Site Erythema (N=1297, 445) | 17 | 21
  Injection Site Induration (N=1297, 446) | 8 | 16
  Any Local (4 month vaccination) (N=1262, 420) | 46 | 54
  Injection Site Tenderness (N=1255, 418) | 37 | 42
  Injection Site Erythema (N=1257, 417) | 19 | 29
  Injection Site Induration (N=1257, 417) | 9 | 17
  Any Local (6 month vaccination) (N=1120, 374) | 41 | 50
  Injection Site Tenderness (N=1106, 372) | 30 | 37
  Injection Site Erythema (N=1104, 370) | 22 | 29
  Injection Site Induration (N=1107, 370) | 9 | 19
  Any Local (12 month vaccination) (N=1102, 355) | 47 | 57
  Injection Site Tenderness (N=1098, 353) | 39 | 50
  Injection Site Erythema (N=1095, 349) | 21 | 30
  Injection Site Induration (N=1095, 351) | 10 | 23
  Any Systemic (2 month vaccination) (N=1313, 451) | 77 | 73
  Rash (N=1296, 446) | 3 | 3
  Change in Eating Habits (N=1289, 446) | 23 | 24
  Sleepiness (N=1297, 447) | 52 | 52
  Persistent crying (N=1299,46) | 42 | 40
  Irritability (N=1300, 446) | 59 | 59
  Vomiting (N=1298, 446) | 10 | 9
  Diarrhea (N=1299, 446) | 16 | 11
  Fever ( ≥ 38°C) (N=1297, 446) | 3 | 2
  Analges.Antipyr.Meds (N=1302, 448) | 66 | 60
  Any Systemic (4 month vaccination) (N=1262, 420) | 65 | 63
  Rash (N=1253, 416) | 3 | 4
  Change in Eating Habits (N=1245, 414) | 18 | 17
  Sleepiness (N=1253, 416) | 38 | 37
  Persistent Crying (N=1254, 417) | 31 | 28
  Irritability (N=1254, 416) | 50 | 48
  Vomiting (N=1254, 416) | 8 | 6
  Diarrhea (N=1255, 416) | 11 | 8
  Fever ( ≥ 38°C) (N=1251, 416) | 4 | 6
  Analges.Antipyr.Meds (N=1254, 416) | 58 | 55
  Any Systemic (6 month vaccination) (N=1120, 374) | 58 | 54
  Rash (N=1101, 367) | 3 | 3
  Change in Eating Habits (N=1094, 367) | 17 | 14
  Sleepiness (N=1104, 367) | 31 | 29
  Persistent Crying (N=1103, 368) | 26 | 20
  Irritability (N=1104, 369) | 46 | 41
  Vomiting (N=1106, 369) | 6 | 4
  Diarrhea (N=1102, 369) | 8 | 6
  Fever ( ≥ 38°C) (N=1108, 368) | 7 | 6
  Analges.Antipyr.Meds (N=1103, 370) | 53 | 49
  Any Systemic (12 month vaccination) (N=1102, 355) | 63 | 62
  Rash (N=1093, 353) | 4 | 5
  Change in Eating Habits (N=1089, 348) | 18 | 16
  Sleepiness (N=1096, 353) | 30 | 29
  Persistent Crying (N=1094, 353) | 28 | 24
  Irritability (N=1094, 354) | 50 | 49
  Vomiting (N=1094, 353) | 5 | 4
  Diarrhea (N=1094, 353) | 12 | 9
  Fever ( ≥ 38°C) (N=1092, 353) | 9 | 8
  Analges.Antipyr.Meds (N=1095, 354) | 49 | 50

4. Secondary Outcome: Number of Subjects Who Reported Unsolicited Adverse Events After Any Vaccination
Description: Safety data with medically attended events were collected throughout the study in the non-detailed safety groups and from Day 8 onwards for the detailed safety groups.
Time Frame: Day 1 (2 months of age) to 18 months of age
Population: Analysis was done on as treated safety population.
Measure: Number; unit: Subjects
Groups:
- MenACWY-CRM197 + Routine Vaccines (All): Infants received one vaccination of MenACWY-CRM197 vaccine at 2, 4, 6 and 12 months of age and one vaccination of routine vaccines (according to the local vaccination schedule) - DTaP: 2, 4, 6, 15 months, IPV: 2, 4, 6, months, Hib: 2, 4, 6, 15 months, Pneumococcal conjugate: 2, 4, 6, 12 months, MMR, Varicella, Hepatitis A: 12 months. HBV and rotavirus vaccines should be administered according to ACIP guidelines during the first year of life.
  Routine vaccines given to subjects in these arms will be consistent with the US ACIP recommended vaccines.
  All (Detailed and Non-Detailed subjects): Detailed - infants who provided reactogenicity and all AEs for 7 days, SAEs and medically attended AEs; Non-Detailed - infants who only provided SAEs and medically attended AEs.
- Routine Vaccines (All): Infants received one vaccination of routine vaccines (according to the local vaccination schedule) - DTaP: 2, 4, 6, 15 months, IPV: 2, 4, 6, months, Hib: 2, 4, 6, 15 months, Pneumococcal conjugate: 2, 4, 6, 12 months, MMR, Varicella, and Hepatitis A: 12 months. HBV and rotavirus vaccines should be administered according to ACIP guidelines during the first year of life.
  Routine vaccines given to subjects in these arms will be consistent with the US ACIP recommended vaccines.
  All (Detailed and Non-Detailed subjects): Detailed - infants who provided reactogenicity and all AEs for 7 days, SAEs and medically attended AEs; Non-Detailed - infants who only provided SAEs and medically attended AEs.
Arm/Group | MenACWY-CRM197 + Routine Vaccines (All) | Routine Vaccines (All)
Number analyzed (Participants) | 5760 | 1968
Subjects
  Any AE | 4848 | 1659
  Any SAE-Total | 354 | 114
  Possibly or Probably Related AEs | 520 | 2
  AEs Leading to Premature Withdrawals | 44 | 8
  Deaths | 7 | 1

ADVERSE EVENTS:
Time Frame: Throughout study period.
Description: Post-injection solicited Adverse Events (AEs) were collected from Days 1-7 after each vaccination in detailed group. Medically attended AEs and Serious AEs were collected throughout the study period. Subjects who terminated early were followed for 6 months post final dose for safety.
Arm/Group | MenACWY-CRM197 + Routine Vaccines (All) | Routine Vaccines (All)
Serious Adverse Events (participants affected / at risk) | 354/5760 | 114/1968
Other Adverse Events (participants affected / at risk) | 4701/5760 | 1600/1968
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY-CRM197 + Routine Vaccines (All) (N=5760) | Routine Vaccines (All) (N=1968)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Idiopathic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0
Mesenteric Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cyanosis (Cardiac disorders) | 2 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 1
Ventricular Tachycardia (Cardiac disorders) | 1 | 0
Anomalous Pulmonary Venous Connection (Congenital, familial and genetic disorders) | 0 | 1
Congenital Absence Of Bile Ducts (Congenital, familial and genetic disorders) | 1 | 0
Congenital Aplastic Anaemia (Congenital, familial and genetic disorders) | 1 | 0
Craniosynostosis (Congenital, familial and genetic disorders) | 1 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 1 | 0
Hamartoma (Congenital, familial and genetic disorders) | 1 | 0
Mitochondrial Enzyme Deficiency (Congenital, familial and genetic disorders) | 1 | 0
Osteognesis Imperfecta (Congenital, familial and genetic disorders) | 1 | 0
Patent Ductus Arteriosus (Congenital, familial and genetic disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 0
Pyloric Stenosis (Congenital, familial and genetic disorders) | 1 | 0
Vitello-Intestinal Duct Remnant (Congenital, familial and genetic disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 3 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Inguinal Hernia (Gastrointestinal disorders) | 2 | 0
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 0 | 1
Intussusception (Gastrointestinal disorders) | 4 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Brain Death (General disorders) | 1 | 0
Hernia (General disorders) | 0 | 1
Pyrexia (General disorders) | 7 | 3
Jaundice (Hepatobiliary disorders) | 1 | 0
Acute Tonsilitis (Infections and infestations) | 1 | 1
Adenovirus Infection (Infections and infestations) | 1 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 1
Ascariasis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial Diarrhoea (Infections and infestations) | 1 | 0
Bacterial Tracheitis (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 64 | 15
Bronchitis (Infections and infestations) | 1 | 3
Bronchopneumonia (Infections and infestations) | 19 | 5
Cellulitis (Infections and infestations) | 5 | 4
Cellulitis Staphylococcal (Infections and infestations) | 1 | 0
Cellulitis Streptococcal (Infections and infestations) | 1 | 0
Chest Wall Abscess (Infections and infestations) | 1 | 0
Croup Infectious (Infections and infestations) | 10 | 5
Diarrhoea Infectious (Infections and infestations) | 1 | 0
Dysentery (Infections and infestations) | 1 | 0
Enterovirus Infection (Infections and infestations) | 1 | 0
Escherichia Urinary Tract Infection (Infections and infestations) | 1 | 2
Exanthema Subitam (Infections and infestations) | 0 | 3
Furuncle (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 20 | 7
Gastroenteritis Rotavirus (Infections and infestations) | 2 | 0
Gastroenteritis Salmonella (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 7 | 3
Genital Abscess (Infections and infestations) | 2 | 0
Groin Abscess (Infections and infestations) | 2 | 0
Haemophilus Bacteraemia (Infections and infestations) | 1 | 0
Hand-Foot-And-Mouth Disease (Infections and infestations) | 10 | 0
Herpangina (Infections and infestations) | 4 | 2
Incision Site Cellulitis (Infections and infestations) | 1 | 0
Infected Cyst (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 4 | 0
Klebsiella Bacteraemia (Infections and infestations) | 1 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0
Lymph Node Abscess (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 1 | 0
Meningitis Enteroviral (Infections and infestations) | 1 | 0
Metapneumovirus Infection (Infections and infestations) | 1 | 0
Otitis Media (Infections and infestations) | 2 | 3
Otitis Media Acute (Infections and infestations) | 1 | 3
Periorbital Cellulitis (Infections and infestations) | 3 | 0
Peritonsillar Abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 31 | 10
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Pneumococcal bacteraemia (Infections and infestations) | 0 | 1
Pneumonia Adenoviral (Infections and infestations) | 1 | 0
Pneumonia Bacterial (Infections and infestations) | 1 | 0
Pneumonia Influenzal (Infections and infestations) | 1 | 0
Pneumonia Primary Atypical (Infections and infestations) | 0 | 1
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 1 | 0
Pneumonia Viral (Infections and infestations) | 3 | 1
Pyelonephritis (Infections and infestations) | 1 | 2
Pyelonephritis Acute (Infections and infestations) | 4 | 0
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 20 | 7
Respiratory Synctial Virus Infection (Infections and infestations) | 4 | 2
Rotavirus Infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 3 | 0
Sinusitis (Infections and infestations) | 0 | 1
Staphylococcal Abscess (Infections and infestations) | 1 | 2
Tonsilitis (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 1
Urachal Abscess (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 28 | 10
Urinary Tract Infection Enterococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 1 | 0
Viral Diarrhoea (Infections and infestations) | 1 | 0
Viral Infection (Infections and infestations) | 4 | 0
Wound Infection (Infections and infestations) | 1 | 0
Accidental Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 5 | 2
Electrical Burn (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Foreign Body (Injury, poisoning and procedural complications) | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 2
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 1
Skull Fracture (Injury, poisoning and procedural complications) | 1 | 1
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram Qt Prolonged (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 18 | 9
Failure To Thrive (Metabolism and nutrition disorders) | 1 | 0
Feeding Disorder (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 2 | 0
Acute Disseminated Encephalomyelitis (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 5 | 3
Encephalitis (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 2 | 0
Febrile Convulsion (Nervous system disorders) | 9 | 6
Hydrocephalus (Nervous system disorders) | 1 | 0
Myoclonic Epilepsy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Breath Holding (Psychiatric disorders) | 1 | 0
Drug Abuse (Psychiatric disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Renal Mass (Renal and urinary disorders) | 0 | 2
Vesicoureteric Reflux (Renal and urinary disorders) | 1 | 0
Balanitis (Reproductive system and breast disorders) | 1 | 0
Scrotal mass (Reproductive system and breast disorders) | 1 | 0
Adenoidal Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Bronchomalacia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 12 | 3
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Status Asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hernia Repair (Surgical and medical procedures) | 1 | 0
Inguinal Hernia Repair (Surgical and medical procedures) | 0 | 1
Angiopathy (Vascular disorders) | 1 | 0
Kawasaki's Disease (Vascular disorders) | 4 | 1
Vasculitis (Vascular disorders) | 1 | 0
Retinal Haemorrhage (Eye disorders) | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 4 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Meningitis Viral (Infections and infestations) | 2 | 0
Subdural Hematoma (Injury, poisoning and procedural complications) | 1 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY-CRM197 + Routine Vaccines (All) (N=5760) | Routine Vaccines (All) (N=1968)
Anaemia (Blood and lymphatic system disorders) | 276 | 94
Conjunctivitis (Eye disorders) | 732 | 234
Constipation (Gastrointestinal disorders) | 275 | 98
Diarrhoea (Gastrointestinal disorders) | 1181 | 356
Teething (Gastrointestinal disorders) | 294 | 106
Vomiting (Gastrointestinal disorders) | 500 | 155
Injection Site Erythema (General disorders) | 519 | 241
Injection Site Induration (General disorders) | 284 | 181
Injection Site Pain (General disorders) | 916 | 338
Irritability (General disorders) | 1146 | 405
Pyrexia (General disorders) | 1239 | 373
Bronchiolitis (Infections and infestations) | 826 | 299
Bronchitis (Infections and infestations) | 446 | 153
Croup Infectious (Infections and infestations) | 284 | 98
Gastroenteritis (Infections and infestations) | 524 | 179
Influenza (Infections and infestations) | 415 | 124
Nasopharyngitits (Infections and infestations) | 751 | 239
Otitis Media (Infections and infestations) | 1579 | 551
Otitis Media Acute (Infections and infestations) | 412 | 154
Pharyngitits (Infections and infestations) | 609 | 208
Sinusitis (Infections and infestations) | 296 | 93
Upper Respiratory Tract Infection (Infections and infestations) | 2358 | 842
Viral Infection (Infections and infestations) | 591 | 175
Crying (Nervous system disorders) | 859 | 277
Somnolence (Nervous system disorders) | 927 | 307
Eating Disorder (Psychiatric disorders) | 593 | 187
Cough (Respiratory, thoracic and mediastinal disorders) | 504 | 171
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 628 | 201
Eczema (Skin and subcutaneous tissue disorders) | 399 | 145
Rash (Skin and subcutaneous tissue disorders) | 307 | 109

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days